CLINICAL TRIAL: NCT00004099
Title: Randomized Phase III Study of Preoperative Chemotherapy Followed by Surgery Versus Surgery Alone in Locally Advanced Gastric Cancer (cT3 and cT4NxM0)
Brief Title: Surgery With or Without Combination Chemotherapy in Treating Patients With Stomach Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-40954; EORTC-40954
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Gastric Cancer
Keywords: stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; intestinal adenocarcinoma of the stomach; diffuse adenocarcinoma of the stomach; mixed adenocarcinoma of the stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Fluorouracil; Leucovorin; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Drug: leucovorin calcium
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if surgery alone or surgery combined with chemotherapy is more effective in treating stomach cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery with or without combination chemotherapy in treating patients who have stage II, stage III, or stage IV stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare overall survival in patients with locally advanced gastric cancer treated with surgery alone or in combination with neoadjuvant cisplatin, leucovorin calcium and fluorouracil.
* Compare these two regimens in terms of the rate of complete resection, time to progression, and morbidity in these patients.
* Evaluate toxicity of and disease response to neoadjuvant chemotherapy in these patients.
* Evaluate quality of life and performance status in these patients pre- and post-surgery and compare quality of life for both regimens.

OUTLINE: This is a randomized, open label, multicenter study. Patients are stratified according to center, primary tumor category (cT3 or cT4), localization of tumor (upper third including cardia II or III vs middle and lower third), gender, and histological subtype (intestinal vs nonintestinal). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive cisplatin IV over 1 hour on days 1, 15, and 29. Patients also receive leucovorin calcium IV over 2 hours followed by fluorouracil IV over 24 hours on days 1, 8, 15, 22, 29, and 36. A second course is administered beginning 2 weeks later in the absence of disease progression or unacceptable toxicity.

Patients undergo resection and lymphadenectomy on days 57-63 of the second course of chemotherapy.

* Arm II: Patients undergo resection and lymphadenectomy within 14 days of randomization.

Quality of life is assessed before randomization, every 3 months for 1 year and at 2 years after randomization.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, then every 3 months thereafter until death.

PROJECTED ACCRUAL: A total of 360 patients (180 per arm) will be accrued for this study over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage II-IV adenocarcinoma of the stomach including cardia carcinoma types II and III

  * Locally resectable disease
  * No distant metastases except M1 lymph nodes
  * No evidence of peritoneal carcinomatosis

    * Free tumor cells in lavage at laparoscopy allowed
* No uncontrolled bleeding of the primary tumor
* No gastric outlet syndrome or complete tumor stenosis that would require total parenteral nutrition

PATIENT CHARACTERISTICS:

Age:

* 18 to 69

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 4,000/mm^3
* Absolute neutrophil count greater than 2,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* Prothrombin rate at least 70%

Renal:

* Creatinine no greater than 1.25 times ULN
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No prior atrial or ventricular arrhythmias
* No prior congestive heart failure
* No myocardial infarction within the past 6 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other prior or concurrent neoplasm except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No active infection
* No allergy to protocol drugs
* No dementia or significantly altered mental status
* No other serious medical condition that would prevent compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No filgrastim (G-CSF) within 48 hours prior to chemotherapy

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics
* No prior stent implantation
* No prior laser therapy

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 1999-07; Primary Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schuhmacher, Study Chair — Technical University of Munich
Locations (18):
- Institut Jules Bordet, Brussels, Belgium
- National Cancer Institute of Egypt, Cairo, Egypt
- Germany (14):
  - Robert Roessle Klinik, Berlin
  - Klinik & Poliklinik fur Strahlentherapie der Universitat zu Koln, Cologne
  - Medizinische Klinik I, Dresden
  - Universitaetsklinik Duesseldorf, Düsseldorf
  - Department of Medicine III, Erlangen
  - Kliniken Essen - Mitte, Essen
  - Evangelisches Bethesda Krankenhaus GmbH, Essen
  - Krankenhaus Nordwest, Frankfurt
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Universitatsklinik - Saarland, Homburg
  - Kreiskrankenhaus Meissen, Meissen
  - Klinikum Rechts Der Isar/Technische Universitaet Muenchen, Munich
  - Westfaelische Wilhelms-Universitaet, Münster
  - Staedtisches Krankenhaus, Solingen
- Academisch Ziekenhuis Maastricht, Maastricht, Netherlands
- Instituto Portugues de Oncologia Centro do Porto, SA, Porto, Portugal

REFERENCES:
- [Result] Schuhmacher C, Gretschel S, Lordick F, Reichardt P, Hohenberger W, Eisenberger CF, Haag C, Mauer ME, Hasan B, Welch J, Ott K, Hoelscher A, Schneider PM, Bechstein W, Wilke H, Lutz MP, Nordlinger B, Van Cutsem E, Siewert JR, Schlag PM. Neoadjuvant chemotherapy compared with surgery alone for locally advanced cancer of the stomach and cardia: European Organisation for Research and Treatment of Cancer randomized trial 40954. J Clin Oncol. 2010 Dec 10;28(35):5210-8. doi: 10.1200/JCO.2009.26.6114. Epub 2010 Nov 8. PMID 21060024
- [Result] Schuhmacher C, Schlag P, Lordick F, et al.: Neoadjuvant chemotherapy versus surgery alone for locally advanced adenocarcinoma of the stomach and cardia: randomized EORTC phase III trial #40954. [Abstract] J Clin Oncol 27 (Suppl 15): A-4510, 2009.